CLINICAL TRIAL: NCT04374708
Title: Gender Identity and Own Body Perception- Implications for the Neurobiology of Gender Dysphoria
Brief Title: Gender Identity and Own Body Perception
Status: Terminated | Type: Observational
Why Stopped: The funding agency, the NICHD, did not make a non-competing continuation award for the fifth and final year of the project and moved the grant into closeout.
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Jamie Feusner, Professor of Psychiatry and Biobehavioral Sciences, University of California, Los Angeles
Other Study IDs: 1R01HD087712-01A1 (NIH)
Record Dates: First submitted 2020-04-19; First posted 2020-05-05 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Gender Dysphoria
MeSH Terms: conditions — Gender Dysphoria | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- trans men: fMRI: body morph test and neurocognitive testing
  Interventions: Diagnostic Test: fMRI
- trans women: fMRI: body morph test and neurocognitive testing
  Interventions: Diagnostic Test: fMRI
- homosexual cisgender men: fMRI: body morph test and neurocognitive testing
  Interventions: Diagnostic Test: fMRI
- homosexual cisgender women: fMRI: body morph test and neurocognitive testing
  Interventions: Diagnostic Test: fMRI
- cisgender women: fMRI: body morph test and neurocognitive testing
  Interventions: Diagnostic Test: fMRI
- cisgender men: fMRI: body morph test and neurocognitive testing
  Interventions: Diagnostic Test: fMRI

INTERVENTIONS:
Diagnostic Test: fMRI — fMRI: body morph test and neurocognitive testing

SUMMARY:
This study will provide valuable information on the neurobiological underpinning of gender dysphoria (GD) and the effects of sex hormones, and promises to uncover functional or structural neural patterns that could predict outcome in terms of body image and quality of life after cross-sex hormone treatment.

DETAILED DESCRIPTION:
The purpose of this study is to understand the neurobiology of gender dysphoria (GD) and the interactions between cross hormone treatment, the brain, and the body phenotype. The investigators also aim to identify pre-treatment neurobiological and other factors to help predict body congruence and quality of life outcomes from hormone treatment. There is mounting interest in gender identity issues worldwide, as requests for gender-confirming treatments have increased in the past 3 decades, and alarmingly high suicide rates have recently been reported in those with GD. Despite this, little is known about neurobiological or other etiological factors contributing to GD or gender incongruence. This study will address a core feature of GD that has been little studied in terms of the neurobiology: the incongruence between perception of self and one's own body.

ELIGIBILITY:
Participants with gender dysphoria (GD)

Inclusion Criteria:

* Females and males from any racial or ethnic background, between the ages of 18 years and 40 years.
* Participants must meet Diagnostic and Statistical Manual-5 criteria for GD (302.85)
* Intelligence quotient (IQ) > 80

Participants with GD

Exclusion Criteria:

* Previous or on-going sex hormone medication
* Previous sex reassignment surgery
* Oral contraceptives
* Participants with GD are not be taking any other psychotropic medication. (No participant will be recommended to discontinue or taper medications for the purpose of participating in the study.)
* Irregular menstrual cycles

Control participants

Inclusion Criteria:

* Females and males from any racial or ethnic background, between the ages of 18 and 40.
* IQ > 80

Control participants

Exclusion Criteria:

* Psychiatric medications
* A score of ≥ 1 standard deviation higher than population norms on the MADRS depression or the Hamilton anxiety scale (HAMA)
* Sex hormone treatment
* Irregular menstrual cycles

Exclusion criteria for all participants:

* Any known chromosomal or hormonal disorder
* Current substance abuse or dependence
* Current neurological disorder or psychiatric disorder
* Pregnancy
* Current major medical disorders that may affect cerebral metabolism such as diabetes or thyroid disorders
* Head trauma associated with loss of consciousness
* HIV positive individuals
* Individuals with ferromagnetic metal implantations or devices. This includes any electronic implants or devices, braces, infusion pumps, aneurysm clips, metal fragments or foreign bodies, metal prostheses, joints, rods or plates
* Visual acuity worse than 20/35 for each eye as determined by Snellen close vision acuity chart. Acuity may be met with corrective lenses

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Investigators will enroll 150 participants between the ages of 18 and 40 (25 trans males; 25 trans females; 25 cis gender females; 25 cis gender males; 25 homosexual males; 25 homosexual females)
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
cerebral networks measured by functional magnetic resonance imaging (fMRI) mediating body perception and association with subjective own-body self-incongruence | Baseline Visit 2 pre hormone treatment
  Own body perception in relation to functional and structural connection
Morphometric differences by sex, gender identity and sexual orientation | Baseline Visit 2 pre hormone treatment
  Cortical thickness, surface area, cortical and subcortical structural volumes and white matter tracts measured by MRI in relation to sex and gender identity and sexual orientation.
Brain activation during own body perception | Baseline Visit 2 pre hormone treatment
  Images of body morph test presented during fMRI scan
Change in cerebral networks measured by functional magnetic resonance imaging (fMRI) mediating body perception and association with subjective own-body self-incongruence | Post hormone treatment. Visit 4 last appt. within 2 yrs of Visit 2.
  Own body perception in relation to functional and structural connection
Change in morphometric differences by sex, gender identity and sexual orientation | Post hormone treatment. Visit 4 last appt. within 2 yrs of Visit 2.
  Cortical thickness, surface area, cortical and subcortical structural volumes and white matter tracts measured by MRI in relation to sex and gender identity and sexual orientation.
Change in brain activation during own body perception | Post hormone treatment. Visit 4 last appt. within 2 yrs of Visit 2.
  Images of body morph test presented during fMRI scan

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No